CLINICAL TRIAL: NCT05881590
Title: Real-world Evidence Feasibility Trial, in Both Community and Hospital-based Settings, for a Technology-enabled Hybrid Service Delivery Model for Pulmonary Rehabilitation: Assessing Patient Uptake and Adherence, and Impact on Patient Outcomes and Service Capacity.
Brief Title: Hybrid Pulmonary Rehabilitation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Aseptika Ltd. (Unknown); So What? Consultancy Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HEMS_2223001
Record Dates: First submitted 2023-04-17; First posted 2023-05-31 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Disease
Keywords: Pulmonary Rehabilitation; hybrid delivery; real-word design; quantitative and qualitative research; health economic analysis
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Intervention Model Description: Real-world study design drawing largely on routinely collected data to compare outcomes for patients recruited to a hybrid pulmonary rehabilitation programme with a propensity matched control group that has previously received standard pulmonary rehabilitation as part of usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid pulmonary rehabilitation (Experimental)
  Interventions: Other: Hybrid pulmonary rehabilitation

INTERVENTIONS:
Other: Hybrid pulmonary rehabilitation — Technology-enabled 8-week pulmonary rehabilitation programme using the Active+me REMOTE App

SUMMARY:
Pulmonary rehabilitation is an exercise and education programme that helps improve breathlessness and quality of life for people living with lung and breathing problems. It improves exercise levels and breathlessness and is a recommended treatment for people with lung diseases and symptoms. Standard pulmonary rehabilitation programmes involve individuals attending group classes at hospitals or community centres, twice a week for 8 weeks. These classes are supervised by physiotherapists. At the moment, there are long waiting times for pulmonary rehabilitation in the NHS.

Some patients may prefer more pulmonary rehabilitation based in their own home. This might be because they find it difficult to travel to classes. Some would like to do more home pulmonary rehabilitation in between supervised classes or continue pulmonary rehabilitation after the 8-week supervised programme. The blending between supervised classes and home pulmonary rehabilitation is known as HYBRID PULMONARY REHABILITATION. Hybrid pulmonary rehabilitation is not being provided routinely in the NHS, but the NHS would like to see it used more as it might help reduce waiting times and give patients more choice on how to access pulmonary rehabilitation.

The study will assess the feasibility of a larger study to provide strong evidence on patients' uptake and adherence to the hybrid programme, and the impact on patients' health outcomes and service delivery. The investigators will also look at what measures would be best to use in a larger study.

The study will recruit up to 100 patients. These individuals will be aged 18 years or older, have respiratory disease and a referral for pulmonary rehabilitation. Individuals with reasons why they cannot exercise will be excluded.

Participants will be provided with an application (App) that can be installed on a mobile phone. This App is called Active+me REMOTE and is made by a company called Aseptika Ltd (www.activ8rlives.com). Active+me REMOTE provides live online, video exercise classes; pre-recorded exercise classes; a walking programme; educational talks; and a care plan personalised for the user.

Data will be collected at the beginning and end of the hybrid pulmonary rehabilitation programme and will include routinely collected data as part of usual care. Additional data will be collected via the App and trial surveys. The investigators will ask staff and patients about the experiences of the new way of delivering rehabilitation and explore how cost effective it is.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) for patients with respiratory disease, e.g. chronic obstructive pulmonary disease (COPD) and bronchiectasis, improves exercise capacity, quality-of-life and provides vital education for condition management. PR is now recommended for all COPD patients (NICE guidelines NG115).

A standard PR programme involves two, in-person, exercise classes per week over a period of 8 weeks after which the patient is discharged to self-care. While retaining some in-person contact, technology could increase access and automate delivery of education and exercise by overcoming shortages of skilled staff. New technology exists to allow the delivery of a hybrid PR programme which may be used to support a move to a remotely delivered service (with patients having the opportunity to attend in-person PR sessions during the programme if they need the motivation or support of an in-person session).

This study will use the UKCA/CE Class I-approved and DTAC-certified Active+me REMOTE App (Aseptika Ltd www.activ8rlives.com). The Active+me App, accessible by patients on their smartphones with Bluetooth or connected medical monitors, includes remote tracking of adherence, symptoms and physiological parameters (where appropriate); live, online video exercise classes; pre-recorded classes; a paced walking programme; an educational programme delivered in bite-sized pieces; and personalised care plans for every patient.

Generally, NICE guidance draws on randomised controlled trials (RCTs) to inform guidelines however RCTs are costly and time consuming for digital healthcare and this delays uptake and adoption by the NHS. New and innovative approaches to obtaining effectiveness evidence for digitally delivered healthcare are urgently needed and new approaches and solutions are being reviewed by NICE. This feasibility study will use a real-world study design drawing on routinely collected data to compare outcomes for patients recruited to a Hybrid PR Intervention with a propensity-matched Control Group that has previously received Standard PR. Additional data will be collected from the Hybrid PR group (via Active+me REMOTE / Trial Surveys) to provide supporting evidence relating to uptake, adherence, clinical outcomes (not routinely recorded in standard practice), and usability/acceptability of the Hybrid PR programme.

Patients with chronic respiratory disease who are referred to the Harefield Pulmonary Rehabilitation Programme will be screened for eligibility to participate in the Hybrid PR Trial. Informed consent will obtained in eligible patients who wish to take part. Recruited participants will follow a hybrid PR programme (Intervention Group). The Control Group will be patients that have previously received a standard pulmonary rehabilitation programme and are matched on specified criteria including age, sex, measure of respiratory disability, index of multiple deprivation, exercise capacity and hospital vs community location.

Following their informed consent the Hybrid PR Intervention Group will attend an onboarding session where a member of the clinical research team will i) download the Active+me REMOTE App onto patients' smartphone (or provide patients without a smartphone, one on which the App is preloaded), and ii) connect the patients' Active+me REMOTE account to the clinical team via a secure clinical portal. The clinician will also assign appropriate monitoring devices (e.g. BP monitor, Inhaler tracker, smart (weight) scale, pulse oximeter, peak flow monitor) to the participant. After saving the participant's details the patient's App dashboard will be displayed and (as required) the clinician will demonstrate exercise/ educational content of the App.

Participants will have a preliminary in-person assessment with a member of the Harefield Pulmonary Rehabilitation Team (as part of routine care). The participant will then follow the 8-week Hybrid PR intervention involving two exercise classes per week. While this is an 8-week programme, this may be extended to up to 12 weeks for some patients (for example, if the patient is not able to attend 2 sessions per week). After completing the Hybrid PR programme, the participant will have a discharge assessment (as part of routine care).

Demographic data from routine medical records and data on service location (i.e. hospital vs community setting) will be collected at baseline for the Hybrid PR Intervention and the Control Group. Data from routine medical records will be collected both at baseline and on completing the Hybrid/Standard PR programme. These data will include measures of exercise capacity; disease knowledge; lower limb function; health-related quality of life; anxiety and depression; and breathlessness. Additional research data collection in the Hybrid PR Group will include:

* a questionnaire at baseline and on completion of the intervention to measure patient activation (i.e. knowledge, skills, and confidence to manage their own health/wellbeing). This will be administered by a member of the clinical research team who will add the information to the Clinical Portal
* A symptoms survey built into the Active+me App, which will be completed daily
* Uptake/adherence to the Hybrid PR programme including number of sessions completed/dropouts; activity adherence; educational adherence; and medication adherence (this will be remotely tracked via the Active+me App).

The study will undertake qualitative interviews/focus groups in staff and patient participants involved in the Hybrid PR Programme.

The eligibility criteria for the interviews/focus groups will be:

i) Hospital staff delivering Hybrid PR via the Active+me REMOTE platform. ii) Patients who have agreed to take part in the Hybrid PR intervention

For the qualitative component, staff will be sent an email invite to participate in a focus group, together with an information sheet and a copy of the consent form. As part of their informed consent for taking part in the Hybrid PR intervention, patient participants will be given the option to agree to take part in the qualitative component. Not all patients who agree to the qualitative component will be invited to take part, instead a purposively selected group with a broad range of characteristics (e.g. age, gender, stage of disease) will be selected.

The qualitative research with staff will explore the experience of delivering the Hybrid PR programme, whether anticipated and unanticipated barriers were overcome, and perceptions of success. Any potential cost savings will be explored. Interviews/focus groups with patient participants will address their experience of the Hybrid PR programme, and the barriers and facilitators to using different components of the blended PR pathway.

This feasibility study will generate evidence to support larger trial to compare effectiveness of a Hybrid PR vs Standard PR delivery model on patient uptake, adherence and outcomes, and service capacity. The aim of the larger trial is to provide definitive evidence to inform clinical guidelines for PR delivery.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 years or older
* Have a grade of 2 - 5 on the MRC Dyspnoea Scale and are referred for pulmonary rehabilitation
* Are willing and have capacity to consent to take part in the trial

Exclusion Criteria:

- contraindications to exercise (e.g. unstable cardiac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Feasibility - patient recruitment rates | 4 months (recruitment rate: 6 patients per week)
  Number of patients recruited within the anticipated recruitment timeframe of the study
Feasibility - recruitment | 4 months
  Frequency of reasons for non-participation
Feasibility - participant retention rates | 6 months [from recruitment start to end of data collection]
  The percentage of participants who do not withdraw from the study once consented
Feasibility - Availability of data for primary and secondary outcomes of a larger definitive trial | At the end of the 8-week intervention
  The percentage of missing data extracted from routine records and trial surveys
Feasibility - success of propensity matching of control group | Baseline
  Similarities in the baseline characteristics of intervention arm and retrospective control group including: age (years); sex (M/F); measure of respiratory disability (Grade 0-4), socioeconomic status (index of multiple deprivation); exercise capacity (incremental shuffle walk test); and hospital vs community setting.
Feasibility - Success of integrating hybrid pulmonary rehabilitation into routine practice | 5-6 months
  Qualitative feedback via focus groups from pulmonary rehabilitation staff teams
Feasibility - patient/staff acceptability of the hybrid pulmonary rehabilitation programme | 5-6 months
  Qualitative feedback via interviews/focus groups from patients/pulmonary rehabilitation staff teams
Feasibility - safety of the hybrid pulmonary rehabilitation programme | 6 months [from recruitment start to end of data collection]
  Number of adverse events recorded in participants

SECONDARY OUTCOMES:
Patient uptake of the hybrid pulmonary rehabilitation programme | At the end of the 8-week intervention
  Proportion of eligible participants that agree to take part in the study Hybrid PR intervention and complete at least one class
Pulmonary rehabilitation class sessions completed | At the end of the 8-week intervention/programme
  Number of pulmonary rehabilitation class sessions completed in the hybrid and standard pulmonary rehabilitation programmes
Drop out rate from pulmonary rehabilitation | At the end of the 8-week intervention/programme
  Number of people who drop out of the hybrid and standard pulmonary rehabilitation programmes
Changes in exercise capacity measures | Change from baseline until the end of the 8-week intervention/programme
  Changes in the incremental shuffle walk test in the hybrid and standard pulmonary rehabilitation programmes
Adherence to the hybrid pulmonary rehabilitation programme (activity adherence) | At the end of the 8-week intervention
  Number of minutes of physical activity per week (using data collected via Active+me REMOTE) and number of steps taken per week (using data collected via Active+me REMOTE)
Adherence to the hybrid pulmonary rehabilitation programme (educational adherence) | At the end of the 8-week intervention
  Number of educational lessons read (using data collected via Active+me REMOTE)
Adherence to the hybrid pulmonary rehabilitation programme (medication adherence) | At the end of the 8-week intervention
  Inhaler preventer usage (using data collected via Active+me REMOTE)
Changes in symptoms | Change from baseline until the end of the 8-week intervention/programme
  Changes in breathlessness scores (using MRC Dyspnoea Scale) in the hybrid and standard pulmonary rehabilitation programmes. The scale ranges from 1 (no respiratory disability) to 5 (almost complete incapacity).
Changes in knowledge, skills, and confidence to manage health and wellbeing | Change from baseline until the end of the 8-week intervention/programme
  Changes in the Patient Activation Measure in the hybrid pulmonary rehabilitation programme
Number of reported symptoms during the hybrid pulmonary rehabilitation programme | Change from baseline until the end of the 8-week intervention/programme
  Descriptive measures (e.g. mean, SD, median, IQR, frequencies) relating to number of symptoms collected via Active+me REMOTE App symptoms survey
Changes in disease knowledge | Change from baseline until the end of the 8-week intervention/programme
  Changes in Lung Information Needs Questionnaire Score in the hybrid and standard pulmonary rehabilitation programmes. The minimum score (low information needs) is 0 and the maximum score (high information needs) is 25.
Changes in lower limb function | Change from baseline until the end of the 8-week intervention/programme
  Changes in Short Physical Performance Battery (and components) in the hybrid and standard pulmonary rehabilitation programmes. The overall score range is 0 to 12, with 0 indicating the lowest physical performance, and scores of 12 indicating the highest performance
Changes in lower limb function | Change from baseline until the end of the 8-week intervention/programme
  Changes in bi-lateral knee extension (1-RM) in the hybrid and standard pulmonary rehabilitation programmes
Changes in health-related quality of life | Change from baseline until the end of the 8-week intervention/programme
  Changes in EQ-5D-5L scores in the hybrid and standard pulmonary rehabilitation programmes
Changes in health-related quality of life | Change from baseline until the end of the 8-week intervention/programme
  Changes in disease-specific quality of scores using COPD Assessment Test in the hybrid and standard pulmonary rehabilitation programmes.
Changes in health-related quality of life | Change from baseline until the end of the 8-week intervention/programme
  Changes in disease-specific quality of scores using Chronic Respiratory Questionnaire in the hybrid and standard pulmonary rehabilitation programmes.
Changes in anxiety measures | Change from baseline until the end of the 8-week intervention/programme
  Changes in Hospital Anxiety and Depression Scale - Anxiety (HADS-A) in the hybrid and standard pulmonary rehabilitation programmes. The scale has 7 items each with a scale of 0-3. The minimum score is 0 and the maximum score is 21 (0-7 = normal, 8-10 = borderline abnormal, and 11 - 21 = abnormal)
Changes in depression measures | Change from baseline until the end of the 8-week intervention/programme
  Changes in Hospital Anxiety and Depression Scale - Depression (HADS-D) in the hybrid and standard pulmonary rehabilitation programmes. The scale has 7 items each with a scale of 0-3. The minimum score is 0 and the maximum score is 21 (0-7 = normal, 8-10 = borderline abnormal, and 11 - 21 = abnormal)
Patient costs | At the end of the 8-week intervention
  Travel costs associated with the hybrid and standard rehabilitation programmes (with distances/time travelled calculated from first 3 letters of participants postcode).
Health care resources - service capacity | At the end of the 8-week intervention
  The number of patients that can be offered pulmonary rehabilitation in the hybrid and standard rehabilitation programmes.
Health care resources - waiting times | At the end of the 8-week intervention
  Patient waiting times (weeks/days) for pulmonary rehabilitation in the hybrid and standard rehabilitation programmes.
Health care resources - health care professionals time | At the end of the 8-week intervention
  Health care professionals time (hours) in delivering he hybrid and standard rehabilitation programmes.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Ball, PhD, BSc, Study Director — Anglia Ruskin University
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust - Harefield Hospital, Harefield, Uxbridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
No IPD sharing plan has been developed